CLINICAL TRIAL: NCT07013903
Title: Effects of Kneipp Hydrotherapy During Inpatient Post-Covid-19 Rehabilitation: A Randomized Controlled Trial
Brief Title: Effects of Hydrotherapy During Post-COVID-19 Rehabilitation
Acronym: HydroCoVital A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Bavarian Health and Food Safety Authority (LGL) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Professor, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HydroCoVital A
Record Dates: First submitted 2025-06-05; First posted 2025-06-10 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Post-COVID / Long-COVID; POST-Covid 19; Post COVID Syndrome; Post-COVID Condition
Keywords: rehabilitation; therapy; Post-COVID; Long COVID; intervention; hydrotherapy; Kneipp; balneotherapy; Post-COVID condition; quality of life
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician that performs the final data analysis is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-COVID Rehabilitation with hydrotherapy (Experimental): Cold water hydrotherapy (5-10 minutes each), twice daily during the 3-week multimodal inpatient rehabilitation program and once daily during the 6-month follow-up period
  Interventions: Other: Standard rehabilitation plus cold water hydrotherapy
- Post-COVID Rehabilitation without hydrotherapy (Active Comparator): 3-week inpatient multimodal inpatient rehabilitation program without hydrotherapy
  Interventions: Other: Standard rehabilitation only

INTERVENTIONS:
Other: Standard rehabilitation plus cold water hydrotherapy — Cold water hydrotherapy (5-10 minutes each), twice daily during the 3-week multimodal inpatient rehabilitation program and once daily during the 6-month follow-up period
  Arms: Post-COVID Rehabilitation with hydrotherapy
Other: Standard rehabilitation only — same rehabilitation program than the experimental group but without hydrotherapy
  Arms: Post-COVID Rehabilitation without hydrotherapy

SUMMARY:
This randomized controlled study evaluates the effects of cold water hydrotherapy as an adjunct to standard rehabilitation in patients with Post-COVID Syndrome. The primary aim is to assess changes in quality of life compared to standard rehabilitation alone.

DETAILED DESCRIPTION:
Patients recovering from Post-COVID Syndrome often experience persistent fatigue, autonomic dysregulation, microcirculatory disturbances, and low-grade inflammation, all of which may hinder their return to full function. Kneipp hydrotherapy-using cold water applications-can address these pathophysiological changes through several mechanisms:

Autonomic regulation: Cold stimuli trigger parasympathetic activation and improve sympathovagal balance, helping to stabilize heart rate variability and reduce symptoms of dysautonomia often seen in Post-COVID.

Enhanced microcirculation: Repeated vasoconstriction and reactive vasodilation promote endothelial function and tissue perfusion, which may alleviate muscle aches, dizziness, and fatigue by improving oxygen and nutrient delivery.

Anti-inflammatory effects: Hydrothermal stimuli have been shown to modulate cytokine profiles, increasing anti-inflammatory mediators and potentially dampening the persistent, low-grade inflammation implicated in Post-COVID pathophysiology.

Musculoskeletal recovery: Thermo-mechanical stimulation relaxes tense muscle fibers, reduces pain perception, and supports gradual increases in physical capacity, all of which are important for overcoming Post-COVID deconditioning.

Taken together, these effects suggest that adjunctive cold water hydrotherapy could accelerate functional recovery, reduce symptom burden, and enhance quality of life in Post-COVID rehabilitation.

Baseline Assessments:

At baseline, demographic data including sex, age, height, and weight will be collected. Participants will report their current main Post-COVID symptoms, which will be categorized into symptom clusters: Fatigue (A), Cognitive (B), and Somatic (C). Smoking history will be assessed, including smoking status (current, former, or never), number of cigarettes per day, years of smoking, and pack-years.

The time (in months) since the COVID-19 infection that led to Post-COVID syndrome will be documented, along with the number of COVID-19 vaccinations received at the time of infection. Employment status will be recorded, distinguishing between full-time or part-time employment, COVID-related work disability, retirement, unemployment, or disability pension.

Comorbidities will be documented across the following categories: cardiovascular, pulmonary, cerebrovascular, metabolic, musculoskeletal, psychiatric, and other conditions. The severity of the acute COVID-19 illness will be assessed using the WHO Clinical Progression Scale, including information on any hospital admission and length of stay (in days).

Pulmonary function testing at baseline (V1) will include FEV₁, FVC, FEV₁/FVC ratio, and total lung capacity (TLC), all expressed as percent predicted. Autonomic function will be evaluated using the Schellong test. Vascular status will be assessed by four-limb blood pressure measurement. Additionally, self-reported work ability and the number of Post-COVID-related sick leave days within the past 12 weeks will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Post-COVID Syndrome (ICD-10 code: U08.9)
* Barthel-Index >80
* Referred to the reference center for Post-COVID rehabilitation
* Owning a smartphone to receive digital questionnaires and to use the measurement app for heart rate variability
* Written informed consent

Exclusion Criteria:

* Existing contraindications for Kneipp hydrotherapy like severe cardiovascular diseases (e.g., decompensated heart failure, unstable angina pectoris, acute myocardial infarction), severe venous diseases (e.g., acute deep vein thrombosis of the leg), severe neurological diseases (e.g., uncontrolled epilepsy)
* Prior regular practice of Kneipp applications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life by Short Form-12 Health Survey (SF-12) | From baseline (Visit 1) to end of inpatient rehabilitation (3 weeks, Visit 2)
  Change in the Short Form-12 physical and mental component summary scores

SECONDARY OUTCOMES:
Fatigue severity by Fatigue Severity Scale | From baseline (Visit 1) to end of inpatient rehabilitation (3 weeks, Visit 2)
  Change in Fatigue Severity Scale score
Sleep quality by Pittsburgh Sleep Quality Index | From baseline (Visit 1) to end of inpatient rehabilitation (3 weeks, Visit 2)
  Change in Pittsburgh Sleep Quality Index score
Health status by EuroQol-5 Dimensions-5 Levels | From baseline (Visit 1) to end of inpatient rehabilitation (3 weeks, Visit 2)
  Change in EuroQol-5 Dimensions-5 Levels questionnaire score
Autonomic function (heart rate variability by photoplethysmography) | Daily during first 3 weeks of rehabilitation (Visit 1 to Visit 2)
  Change in heart rate variability (root mean square of successive differences) measured by Kyto 2935 via photoplethysmography
Resting blood pressure (systolic and diastolic) | Daily during first 3 weeks of rehabilitation (Visit 1 to Visit 2)
  Change in morning resting systolic and diastolic blood pressure
Post-COVID work-absence days | From baseline (Visit 1) to 3 months (Visit 3) and to 6 months (Visit 4)
  Number of days of work absence due to Post-COVID-19 symptoms during the past 12-weeks
Long-term quality of life by Short Form-12 | From baseline (Visit 1) to 3 months (Visit 3) and to 6 months (Visit 4)
  Change in Short Form-12 scores at follow-up
Long-term fatigue by Fatigue Severity Scale | From baseline (Visit 1) to 3 months (Visit 3) and to 6 months (Visit 4)
  Change in Fatigue Severity Scale score at follow-up
Adherence to hydrotherapy | During the 3-week intervention phase (up to Visit 2) and over the 6-month follow-up period (to Visit 4)
  Proportion of prescribed hydrotherapy applications in the intervention group performed, as recorded in diary or app.
  Short-term Adherence: During the 3-week intervention phase, patients are considered "adherent" if they perform at least one hydrotherapy session per day on at least 75% of study days. We will compare health improvements between high-adherence and low-adherence participants.
  Long-term Adherence and Effects: Over the 3- and 6-month follow-up, "adherent" patients are those who continue self-administered hydrotherapy at least four times per week on at least 75% of follow-up weeks. We will assess whether these patients sustain greater gains in quality of life.
Adverse events recording | From start of intervention (Visit 1) through end of study (Visit 4, 6-month follow-up)
  Number and severity of adverse events related to Kneipp hydrotherapy
Long-term heart rate variability changes (HRV) | From baseline (Visit 1) to 3 months (Visit 3) and to 6 months (Visit 4)
  Change in heart rate variability parameters (root mean square of successive differences) measured by photoplethysmography. At follow-up visits patients will measure HRV for 7 consecutive days
Post-exertional malaise severity | From baseline (Visit 1) to 6-month (Visit 4) follow-up
  Change in Post-Exertional Malaise score measured by the DePaul Symptom Questionnaire-Post-Exertional Malaise
Daily well-being documentation | Daily throughout the intervention and 6 months follow-up phase (Visit 1 to Visit 4)
  Self-reported daily well-being recorded via digital diary on a scale from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Rembert Koczulla, MD, Principal Investigator — Schön Klinik Berchtesgadener Land
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No